CLINICAL TRIAL: NCT05079542
Title: Randomized Controlled Clinical Trial of BLT Implants Used for Immediate vs Early Placement and Restored With Lithium-disilicate Glass Ceramic or Sintered Zirconia Crowns on Titanium Bonding Bases.
Brief Title: RCT of BLT Implants Used for Immediate vs Early Placement, Restored With Ceramic Crowns on Titanium Bonding Bases.
Acronym: BLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Dr. med. dent. Malin Strasding, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-117
Record Dates: First submitted 2021-03-17; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Tooth Loss; Dental Implant, Single-tooth
Keywords: immediate implant placement; delayed implant placement; all-ceramic crown; monolithic restoration; titanium base
MeSH Terms: conditions — Tooth Loss | interventions — zirconium oxide

STUDY DESIGN:
Intervention Model Description: In the first phase, participants are randomized to receive implants either immediately or 8 weeks after tooth extraction. In a second phase, participants receive either a restoration out of one material or another, this also being randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immediate implant placement (Experimental): Implant is placed immediately after tooth extraction.
  Interventions: Procedure: Timepoint of Implant placement of Bonelevel tapered implants
- Delayed implant placement (Active Comparator): Implant is placed 8 weeks after tooth extraction.
  Interventions: Procedure: Timepoint of Implant placement of Bonelevel tapered implants
- Lithium disilicate crown (Experimental): Crown out of Lithiumdisilicate is inserted onto the implant.
  Interventions: Combination Product: Material for tooth restoration - Lithiumdisilicate glass ceramic or zirconia
- Zirconia Crown (Active Comparator): Crown out of Zirconia is inserted onto the implant.
  Interventions: Combination Product: Material for tooth restoration - Lithiumdisilicate glass ceramic or zirconia

INTERVENTIONS:
Procedure: Timepoint of Implant placement of Bonelevel tapered implants — Implant surgery on different time points
  Arms: Delayed implant placement; Immediate implant placement
Combination Product: Material for tooth restoration - Lithiumdisilicate glass ceramic or zirconia — Tooth restoration with a certain material
  Arms: Lithium disilicate crown; Zirconia Crown

SUMMARY:
The purpose of this study is to assess the outcome of a new bone level tapered implant when inserted either following an immediate placement protocol or an early placement approach and restored with single crowns out of two different ceramic materials adhesively cemented on a titanium bonding base.

ELIGIBILITY:
Inclusion Criteria:

Subjects must require extraction and replacement of a tooth in the maxillary or mandibular anterior or premolar region with an implant reconstruction.

* ≥22 years of age
* Patient in a good general health
* Adequate bone quality and quantity for one-stage implant placement
* Patient with physical status PS1 and PS2 (according to Physical Status Classification System of the American Society of Anesthesiologists; Attachment 5)
* Adequate bone height of at least 1mm longer than the length of the study implant
* Capable of providing written informed consent.
* Obtained informed consent from the patient and committed to the study and the required follow-up visits.

Exclusion Criteria:

* Patients with a high lip line / smile line

  * Thin mucosal biotype
  * Anatomically not sufficient bone volume or height at implant site to achieve primary stability of the implant
  * Pronounced esthetic expectations
  * Lack of keratinized mucosa at implant site (< 2mm oral and buccal)
  * Women of childbearing potential with a positive urine pregnancy test
  * Patients with inadequate oral hygiene or persistent intraoral infection
  * Smokers exceeding 10 cigarettes / day, or equivalent; patients chewing tobacco
  * Severe bruxism or clenching habits
  * Presence a systemic disease or allergy (e.g. conditions requiring chronic routine prophylactic use of antibiotics or prolonged use of steroids, history of rheumatic heart disease, bacterial endocarditis, cardiac vascular anomalies, prosthetic joint replacements, etc.)
  * Presence or history of receiving intravenous or subcutaneous antiresorptive agents, such as bisphosphonates
  * Presence of mucosal diseases (e.g. erosive lichen planus) in the localized area around the study implant
  * Patients with history of renal failure, bleeding disorders, metabolic bone disorder, uncontrolled endocrine disorders, HIV infection, leucocyte dysfunction and deficiencies, neoplastic disease requiring the use of radiation or chemotherapy, etc.
  * Patients with alcohol or drug abuse
  * Participation in any other clinical trial (drug or device) less that 30 days before implant insertion

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 5 years
  Survival of the implant
Survival of the reconstructions | 5 years
  Survival of prosthetic reconstruction

SECONDARY OUTCOMES:
Mesial and distal bone levels | 5 years
  Peri-implant bone level changes
ISQ values | 3 months
  Measurement of ISQ values during implant surgery and at insertion of crown
Soft tissue volume | 5 years
  Intra-oral digital scans with volumetric software will be used for the soft tissue volume measurements.
Technical and biological outcomes of the restorations | 5 years
  Presence of fractures/chipping, retention loss, screw loosening
Recording the need of GBR procedures | 8 weeks
  Need of GBR procedure or not during surgery